CLINICAL TRIAL: NCT01784588
Title: A Prospective, Non-Randomized, Parallel Cohort, Multi-center Study of the Solyx™ Single Incision Sling System vs. the Obtryx™ II Sling System for the Treatment of Women With Stress Urinary Incontinence
Brief Title: Post Market Study Of Single Incision Sling Versus Transobturator Sling for Stress Urinary Incontinence
Acronym: Solyx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U9915-Solyx
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solyx Single Incision Sling System (Active Comparator): Solyx Single Incision Sling System
  Interventions: Device: Solyx Single Incision Sling System
- Obtryx II Sling System (Active Comparator): Obtryx II Sling System
  Interventions: Device: Obtryx II Sling System

INTERVENTIONS:
Device: Solyx Single Incision Sling System — Solyx Single Incision Sling System
  Arms: Solyx Single Incision Sling System
Device: Obtryx II Sling System — Standard outside-in transobturator sling
  Arms: Obtryx II Sling System

SUMMARY:
The purpose of this research study is to compare the treatment device (Solyx) to a different mesh sling or control device (Obtryx II) for the treatment of symptoms for Stress Urinary Incontinence (SUI). Safety information and patient outcomes will be collected for three (3) years and evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 years of age
2. Willing and able to comply with the study procedures and provide written informed consent to participate in the study (subject or legal representative)
3. Diagnosed with predominant SUI confirmed by positive cough stress test during the protocol required bladder fill procedure (see manual of operations)
4. Confirmed SUI is greater than urge incontinence with the Medical Epidemiologic Social Aspect (MESA) questionnaire
5. Cystometric capacity ≥ 300 cc
6. Post-void residual (PVR) of ≤ 150 cc
7. Medically approved for general, regional or monitored anesthesia

Exclusion Criteria:

1. Subjects who are pregnant, lactating, or planning future pregnancies
2. Subjects with a chief complaint of overactive bladder
3. Subjects with a pattern of recurrent urinary tract infections, defined as ≥ 2 culture-proven urinary tract infections during a 6-month period prior to surgery or ≥ 3 in a 12-month period
4. Subjects with previous surgical procedures for SUI including bulking, urethral sling, bone anchor, Burch procedure, pubo-vaginal sling, and Marshall-Marchetti-Krantz (MMK) procedure. Excluding Kelly plication, Botox, anterior repair, or Inter-Stim
5. Subjects with prior pelvic organ prolapse surgery who experienced mesh complications
6. Subjects with previous radiation therapy to the pelvis
7. Subjects with known or suspected hypersensitivity to polypropylene mesh
8. Subjects with any of the following confounding conditions:

   1. Neurogenic bladder
   2. Urethral stricture and bladder neck contracture
   3. Bladder stones or tumors
   4. Urinary tract fistula or diverticula
   5. Pathology which would compromise implant placement including subjects currently taking anticoagulation therapy
   6. Pathology that would limit blood supply or infections that would compromise healing including chemotherapy, systemic steroids and systemic immunosuppressants
9. Subjects with diabetes and an A1c ≥ 7%
10. Non-English speaking subjects
11. Subjects who have participated in an investigational study (medical device or drug) within 30 days of study entry that may impact analysis of this device or have previously participated in the current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2013-06; Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda White, MD, Principal Investigator — University of Texas; Joseph Schaffer, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (23):
- United States (22):
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Scripps Clinic Carmel Valley, San Diego, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Physicians Regional Healthcare, Naples, Florida
  - Cherokee Women's Health Specialist, Canton, Georgia
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - St Alexius Medical Center, Bismarck, North Dakota
  - Genesis Healthcare System, Zanesville, Ohio
  - Center for Pelvic Health, Franklin, Tennessee
  - University of Texas Southwestern, Austin, Texas
  - University of Texas, Southwestern, Dallas, Texas
  - Baylor University Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Las Colinas OBGYN, Irving, Texas
  - MacArthur OB/GYN Management, LLC, Irving, Texas
  - Kyle P. McMorries, MD, Nacogdoches, Texas
  - Permian Research Foundation, Odessa, Texas
  - Valley Medical Center, Covington, Washington
- Cabrini Medical Centre, Malvern, Australia

REFERENCES:
- [Derived] White AB, Anger JT, Eilber K, Kahn BS, Gonzalez RR, Rosamilia A. Female Sexual Function following Sling Surgery: A Prospective Parallel Cohort, Multi-Center Study of the Solyx Single Incision Sling System versus the Obtryx II Sling System. J Urol. 2021 Sep;206(3):696-705. doi: 10.1097/JU.0000000000001830. Epub 2021 May 6. PMID 33955778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment began on August 1, 2013 and was completed on December 23, 2014.
Period: Overall Study
Arm/Group | Solyx Single Incision Sling System | Obtryx II Sling System
Started | 141 | 140
Completed | 104 | 108
Not Completed | 37 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Solyx Single Incision Sling System | Obtryx II Sling System | Total
Number analyzed (Participants) | 141 | 140 | 281
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (11.6) | 48.9 (11.7) | 49.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 140 | 281
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 35 | 49
  Not Hispanic or Latino | 127 | 105 | 232
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 124 | 123 | 247
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 123 | 140 | 263
  Australia | 18 | 0 | 18
Body Mass Index [Mean (Standard Deviation); unit: lb/in^2] | 29.6 (7.3) | 29.7 (6.3) | 29.6 (6.8)
Smoking Status [Count of Participants; unit: Participants]
  Never | 101 | 88 | 189
  Current | 13 | 22 | 35
  Previous | 27 | 30 | 57
  Unknown | 0 | 0 | 0
Diabetes [Count of Participants; unit: Participants]
  None | 136 | 128 | 264
  Insulin Controlled | 2 | 2 | 4
  Oral Agent Controlled | 2 | 6 | 8
  Diet Controlled | 1 | 4 | 5
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 72 | 80 | 152
  Perimenopausal | 16 | 12 | 28
  Postmenopausal | 53 | 48 | 101
Current Hormone Replacement Therapy (HRT) [Count of Participants; unit: Participants]
  None | 110 | 120 | 230
  Oral Estrogen | 11 | 5 | 16
  Vaginal Estrogen | 11 | 8 | 19
  Combination Replacement Therapy | 7 | 3 | 10
  Transdermal Estrogen | 1 | 0 | 1
  Other | 1 | 4 | 5
Hysterectomy [Count of Participants; unit: Participants]
  None | 101 | 106 | 207
  Vaginal | 13 | 19 | 32
  Laparotomy | 9 | 7 | 16
  Laparoscopy | 9 | 3 | 12
  Laparoscopic Assisted Vaginal | 7 | 3 | 10
  Robotic | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Meeting Definition of Treatment Success at 36 Months, by a Composite of Objective and Subjective Measures
Description: An assessment of improvement in stress urinary incontinence at 36 months, by a composite of objective (negative cough stress test with protocol required bladder fill procedure) and subjective measures (subject self reported improvement in their condition, through the Patient Global Impression of Improvement (PGI-I)). The PGI-I scale rates the patient's improvement or worsening of SUI symptoms relative to baseline. The scale is as follows: 1 - Very much better; 2 - Much better; 3 - A little better; 4 - No change' 5 - A little worse; 6 - Much worse; 7 - Very much worse, with the unit of measure being scores on a scale (lower scores indicate a more positive impression of change). Subjects met the definition of treatment success at 36 months if they had an answer of "No" to the item "Direct observation of urine loss with cough provocation" and an Improvement per the PGI-I (a response of "A little better", "Much better", or "Very much better").
Time Frame: Data presented is for 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Solyx Single Incision Sling System | Obtryx II Sling System
Number analyzed (Participants) | 104 | 108
Participants | 94 | 96
Statistical Analysis 1: Comparison: Solyx Single Incision Sling System vs Obtryx II Sling System; Available Cases Only - Intent-to-Treat; Test type: Non-Inferiority — Non-inferiority (NI) was demonstrated if the entire confidence interval was above -15% at 36 months. The sample size was estimated under the assumption that the proportion of subjects with treatment success is 85% for each of Solyx and Obtryx. For a (one-sided) type I error rate of 0.05, 194 subjects (97 per arm) are needed to have 90% power to demonstrate non-inferiority of Solyx with a NI margin of 15%; Non-inferiority was evaluated using a two-sided 90% confidence interval (CI) for the treatment difference (SIS minus TMUS). The CI was calculated based on the pooling of treatment differences across propensity score strata for a binary endpoint; Adjusted Difference in Percentages = -0.4, 90% CI 2-sided [-8.2 to 7.4]
Statistical Analysis 2: Comparison: Solyx Single Incision Sling System vs Obtryx II Sling System; Available Cases Only - Intent-to-Treat; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; [p-value comment as in outcome 1, analysis 1]; Unadjusted Treatment Difference (%) = 1.5, 90% CI 2-sided [-5.4 to 8.4]

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | Solyx Single Incision Sling System | Obtryx II Sling System
All-Cause Mortality (participants affected / at risk) | 0/141 | 1/140
Serious Adverse Events (participants affected / at risk) | 1/141 | 1/140
Other Adverse Events (participants affected / at risk) | 14/141 | 21/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solyx Single Incision Sling System (N=141) | Obtryx II Sling System (N=140)
Device Extrusion (General disorders) | 1 (1) | 1 (1) — Mesh Extrusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solyx Single Incision Sling System (N=141) | Obtryx II Sling System (N=140)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atonic urinary bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fungal Infection (Infections and infestations) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Mixed incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Sensation of pressure (General disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (2)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 3 (3)
Urinary retention (Renal and urinary disorders) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (9)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Device extrusion (General disorders) | 3 (3) | 5 (5) — Mesh extrusion
Medical device site reaction (General disorders) | 0 (0) | 1 (1) — Mesh exposure
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Boston Scientific Corporation (BSC) for review at least 60 days in advance of submission for publication or presentation to a publisher or other third party. BSC reserves the right to delete any Confidential Information or other proprietary information of BSC (including trade secrets but not including Results) from the proposed publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT01784588/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/88/NCT01784588/SAP_001.pdf